CLINICAL TRIAL: NCT06915493
Title: Blood Glucose Levels in Children During Anesthesia: Incidence of Hypoglycemia During Anesthesia Induction and Its Relationship to Preoperative Fasting
Brief Title: Blood Glucose Levels in Children During Anesthesia
Status: Completed | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Principal Investigator, Thorunn Scheving Eliasdottir, Academic chair, Associate Professor, Landspitali University Hospital
Other Study IDs: 47/2023
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Fasting
Keywords: Pediatrics; Children; General anesthesia; Preoperative fasting; Fasting blood glucose; Hypoglycemia
MeSH Terms: conditions — Fasting; Hypoglycemia | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Capillary blood sample glucose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: General Anesthesia — Blood glucose measurements during general anesthesia

SUMMARY:
This cross-sectional study aims to investigate blood glucose levels in children during general anesthesia and explore the incidence of hypoglycemia after anesthesia induction in relation to preoperative fasting.

Blood glucose will be measured following anesthesia induction and prior to discontinuing the administration of the anesthetic agent.

DETAILED DESCRIPTION:
This cross-sectional study aims to investigate blood glucose levels in children < 18 years during general anesthesia, and explore the incidence of hypoglycemia after anesthesia induction in relation to preoperative fasting.

The purpose is to evaluate whether guidelines for shortening the preoperative fasting period of children at our hospital have resulted in a shorter fasting duration and prevalence of low blood glucose levels during anesthesia induction. Also to shed light on blood glucose levels during general anesthesia and its correlation with intravenous fluid management and administration of steroidal anti-emetics.

Blood glucose sampling will be obtained and measured following anesthesia induction and prior to discontinuing the anesthetic agent. If general anesthesia lasts longer than one hour, additional blood glucose analysis will be conducted one hour after the first measurement.

ELIGIBILITY:
Inclusion Criteria:

Children under 18 years of age who undergo intervention under general anesthesia. The parent or guardian understands and speaks Icelandic.

Exclusion Criteria:

Coexisting disease or treatment that may affect fasting blood glucose level; Preoperative intravenous fluid administration; Beta-blockers; Insulin and corticosteroids, endocrine disorders, acute pain, and emergency interventions.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Convenience sample of children undergoing elective intervention under general anesthesia at Landspítali, the University Hospital of Iceland.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Serum blood glucose level | Immediately/within five minutes after anesthesia induction and prior to discontinuing the anesthesia administration.
  Blood glucose sampling and measured during general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Thorunn S Eliasdottir, PhD, Principal Investigator — Landspitali, the University Hospital of Iceland and University of Iceland
Locations (1):
- Anesthesia Department Landspitali UH, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 2025 - December 2026